CLINICAL TRIAL: NCT01747798
Title: A Pilot Trial to Evaluate the Feasibility Auranofin (Ridaura®) for Asymptomatic Patients With First-Recurrence Epithelial Ovarian Cancer
Brief Title: Auranofin in Treating Patients With Recurrent Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1162; NCI-2012-02207 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-16; First posted 2012-12-12 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2018-10

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Auranofin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (auranofin) (Experimental): Patients receive auranofin PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: auranofin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: auranofin — Given PO
  Other Names: Ridaura
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies auranofin in treating patients with epithelial ovarian, primary peritoneal, or fallopian tube cancer. Immunosuppressive therapy, such as auranofin, may be an effective treatment for epithelial ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the feasibility of conducting a 10-patient pilot study in asymptomatic ovarian cancer patients with cancer antigen (CA 125) elevation.

SECONDARY OBJECTIVES:

I. To explore whether oral gold therapy either stabilizes or lowers the CA 125 level and maintains patients in an asymptomatic state and to provide descriptive data on tumor response and duration of response.

II. To acquire qualitative data on patients' perceptions of learning of CA 125 elevation.

III. To explore whether immunohistochemical staining for PKC iota expression in resected tumor samples appears to be associated with clinical outcomes with auranofin.

OUTLINE:

Patients receive auranofin orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of epithelial ovarian, primary peritoneal, or fallopian cancer from any previous time point
* Completion of initial therapy of epithelial ovarian, primary peritoneal, or fallopian cancer from any previous time point (includes completion of surgery and/or followed by post-operative chemotherapy including maintenance) with no subsequent treatment for progressive disease
* An increase in serum CA 125 level, as defined as follows: 1) normalization of the CA 125 during first-line chemotherapy followed by an increase of >= 100 units/mL; OR 2) normalization of the CA 125 during first-line chemotherapy followed by a doubling of the CA 125 beyond the upper limit of normal with a confirmatory measurement within a period of 4 weeks or less that shows the same or higher CA 125 level
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500
* Platelets (PLT) >= 100,000
* Hemoglobin (HgB) > 9.0 g/dL
* Bilirubin < 1.5 x upper limit of normal (ULN)
* Creatinine within institutional normal limits
* Negative urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willingness to be interviewed by telephone about CA 125 elevation
* Able to provide informed written consent
* Willing to provide tissue blocks for correlative research purposes (please note that if tissue blocks are unavailable, the patient will still be eligible provided they meet all other eligibility criteria)

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease, which in the judgment of the treating oncologist, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Symptoms (other than anxiety, depression, or other psychological symptoms) that, in the opinion, of the treating oncologist are a direct result of cancer recurrence; (examples of symptoms that would preclude enrollment include unintentional weight loss and new abdominal pain)
* Receiving any other prescribed therapy treatment for ovarian cancer
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2015-04-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a 10-patient pilot study in asymptomatic ovarian cancer patients using CA 125 elevation | Up to 2 years
  To demonstrate the feasibility of conducting a 10-patient pilot study in asymptomatic ovarian cancer patients with CA 125 elevation. This study could potentially serve as a paradigm to investigate agents that might eventually be used as maintenance therapy in patients at high risk for recurrent disease.

SECONDARY OUTCOMES:
Immunohistochemical staining for PKCt expression in resected tumor samples with Auranofin | up to 2 years
  To explore whether immunohistochemical staining for PKCt expression in resected tumor samples appears to be associated with clinical outcomes with Auranofin.
Patients' perceptions of learning of CA 125 elevation | up to 2 years
Oral gold therapy influence on the CA 125 levels | 2 years
  To explore whether oral gold therapy either stabilizes or lowers the CA 125 level and maintains patients in an asymptomatic state and to provide descriptive data on tumor response and duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Rousselle B, Massot A, Privat M, Dondaine L, Trommenschlager A, Bouyer F, Bayardon J, Ghiringhelli F, Bettaieb A, Goze C, Paul C, Malacea-Kabbara R, Bodio E. Conception and Evaluation of Fluorescent Phosphine-Gold Complexes: From Synthesis to in vivo Investigations. ChemMedChem. 2022 Jun 3;17(11):e202100773. doi: 10.1002/cmdc.202100773. Epub 2022 Mar 29. PMID 35254001